CLINICAL TRIAL: NCT06683989
Title: Investigating the Effects of Pilates Exercises on Gait Parameters in Pregnant Women: A Randomized Controlled Trial
Brief Title: Effects of Pilates Exercises on Gait in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcan Suicmez (Other)
Responsible Party: Sponsor-Investigator, Selcan Suicmez, Sub-Investigator, Ankara Medipol University
Organization: Ankara Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AnkaraMedipolU-FTR-2024-124
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy; Gait Analysis; Pain
Keywords: pregnancy; pilates training; gait analysis; posture; pain
MeSH Terms: conditions — Pain | interventions — Exercise Movement Techniques; Prenatal Care

STUDY DESIGN:
Intervention Model Description: Our randomized controlled trial divided the participants into a Pilates group (PG) and a control group (CG). Pilates exercises were applied to PG, while CG was given a prenatal care program.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Both the statistical analyst and the evaluator were blind to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pilates group (Experimental): The Pilates exercise program will be conducted for eight weeks, two days per week.
  Interventions: Other: Pilates training
- Control group (Experimental): Regular prenatal care for participants in the CG included standard nursing and medical treatments. Ergonomics information was provided to participants. No exercise regimen was prescribed.
  Interventions: Other: Prenatal care

INTERVENTIONS:
Other: Pilates training — One hour of Pilates training was conducted for eight weeks, two days a week. Every training session was carried out by a certified and experienced physiotherapist from the Australian Institute of Pilates and Physiotherapy. The one-hour session was structured as a warm-up, a cool-down, and Pilates exercises.
  Arms: Pilates group
Other: Prenatal care — Regular prenatal care for participants in the CG included standard nursing and medical treatments.
  Arms: Control group

SUMMARY:
The goal of this interventional study is to investigate how the gait parameters, pain, and posture of women who perform Pilates exercises during pregnancy are affected. This research targets pregnant women without any medical or obstetric complications who are experiencing physiological changes associated with pregnancy.

The main questions it aims to answer are:

Do Pilates exercises influence gait parameters in pregnant women? Does participation in Pilates improve pain and other functional parameters during pregnancy?

Participants will:

Undergo assessments of gait and related parameters. Participate in a Pilates exercise program tailored to their trimester. Provide feedback on pain and overall physical wellness during the study period.

DETAILED DESCRIPTION:
Pregnancy is a physiological process that begins with fertilization and lasts until birth. The pregnancy period typically spans approximately 40 weeks and is divided into three trimesters, each lasting three months. During this process, various critical anatomical, physiological, psychological, and social changes occur in the mother to meet fetal and maternal needs. If the mother's body cannot adequately adapt to these changes, potential health issues that may arise could threaten the health of both mother and fetus.

Pregnancy is a substantial load on the human body, particularly the musculoskeletal system. Pregnancy-related changes in the center of gravity create mechanical stress on the body, accompanied by hormonal changes, increased joint laxity, body weight gain, postural changes, and alterations in the abdominal and pelvic regions. These changes may contribute to postural adaptations, dysfunctions in the lumbar and pelvic regions, and weakening of abdominal muscles.

Regular physical activity significantly benefits pregnant women classified as low-risk with no medical or obstetric complications. Therefore, increasing physical activity levels and regular exercise during pregnancy are recommended in guidelines from the American College of Obstetricians and Gynecologists on physical activity and exercise during pregnancy and the postpartum period. The benefits of regular physical activity and exercise during pregnancy include maintaining and improving physical fitness, preventing excessive gestational weight gain, reducing the risk of preeclampsia and preterm birth, lowering the prevalence of back pain, improving sleep quality, reducing anxiety and depressive symptoms, and enhancing health perception and body image. Based on the results of systematic reviews, regular physical activity and exercise during pregnancy are known to reduce the risk of GDM by 38%, preeclampsia by 41%, gestational hypertension by 39%, macrosomia by 39%, and prenatal depression by 67%. Because of these beneficial effects, it is recommended that pregnant women engage in moderate-intensity aerobic exercise for at least 30 minutes a day, five days a week. However, only about 15% of pregnant women meet the minimum physical activity recommendations (at least 150 minutes of moderate-intensity physical activity per week).

Pilates is an exercise method developed by Joseph Hubertus Pilates that activates all muscular functions of the body, particularly core muscles, increases the endurance, flexibility, and strength of body muscles, and improves balance systems while also enhancing dynamic postural control. Joseph Pilates developed over 600 exercises suitable for all levels and types, with the primary goal of strengthening the core muscles, also known as the "powerhouse" in Pilates, which includes the multifidus, transversus abdominis, pelvic floor, and diaphragm muscles. His aim was to enhance stabilization and distribute the strength generated by these muscles throughout the body, improving the strength, endurance, and flexibility of all muscles, ligaments, and fascia for overall body health. When performed correctly, Pilates exercises enhance physical health and support mental and social well-being.

Due to their training, physiotherapists create personalized exercise programs tailored to each patient, considering the type, intensity, and duration of the activity to prevent potential risks to both the mother and fetus. The stage of pregnancy is crucial in determining these parameters. Pregnancy exercise training programs consist of three phases: warm-up, main exercise, and cool-down phases. These programs are specifically tailored based on a comprehensive biopsychosocial assessment of each individual's needs.

Craig Phillips, a physiotherapist and former ballet dancer, led the foundation of the Australian Physiotherapy and Pilates Institute (APPI) by modifying Pilates exercises to align with body biomechanics. This led to the development of clinical Pilates, now practiced by physiotherapists to ensure scientifically-based, biomechanics-focused Pilates programs suited for pregnant women.

Clinical Pilates positively affects both maternal health and fetal well-being, helping mothers feel more at ease and at peace. Moreover, studies report that online Pilates exercises reduce depression, anxiety, and fear of childbirth in pregnant women. In addition to inner peace and calmness, clinical Pilates is a beneficial technique for achieving breath control, improving spinal stabilization, enhancing pelvic floor control, and promoting proper posture, making it an ideal exercise form for pregnancy.

During pregnancy, clinical Pilates helps increase muscle tone, leading to elongation of the spine. As the spine becomes more flexible, the rib cage elevates, providing more space for fetal development. This increased space not only allows for more manageable fetal growth but also reduces symptoms such as back pain. Stronger muscles and improved physical fitness enhance coordination and balance. Practicing Pilates daily can also increase daily energy levels in pregnant women. Clinical Pilates facilitates proper blood flow, supports fetal nutrition, and provides relaxation for the mother without diverting blood away from the fetus. It aids in maintaining balance, enhances range of motion, and promotes flexibility and strength. The sense of accomplishment from time invested in self-care brings joy and satisfaction, empowering mothers to adapt to temporary physical changes during pregnancy, moving freely and confidently. After pregnancy, clinical Pilates also aids in returning to normal physical health.

Research has shown that the changes experienced during pregnancy can alter gait mechanics, increasing the risk of falling. Studies evaluating gait biomechanics in pregnancy report decreased walking speed, step length, and cadence, with an increase in the double support phase. Blaszczyk and colleagues suggest this change results primarily from weight gain and balance concerns during pregnancy. Another study found increased ankle moments and reduced gluteus maximus activation during walking in pregnant women. The enlargement and forward displacement of the uterus results in a shift in the center of gravity, leading to postural and musculoskeletal changes. Pregnant women may modify their gait parameters to adapt to these changes and maintain balance.

Given the changes that occur during pregnancy and the beneficial effects of Pilates on body systems, investigating the effect of Pilates on gait in pregnant women is warranted. Therefore, this study aims to examine the effects of Pilates exercises on pain and gait parameters in pregnant women.

Our hypotheses are as follows:

H0: Pilates exercises do not affect gait parameters in pregnant women. H1: Pilates exercises affect at least one of the gait parameters in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous and singleton pregnancy was defined as being between 20 and 35
* Being at least in the 16th week of pregnancy

Exclusion Criteria:

* Multiple pregnancies
* Heart and lung problems
* All situations in which exercise is contraindicated during pregnancy
* Participation in different activity programs

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 33 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Gait Analysis | 5 minutes
  Gait parameters will be assessed via the G-Walk. The G-Walk is a device that is worn on the waist via an elastic belt. The G-Walk is built with a triaxial accelerometer 16 bit/axes with multiple sensitivity, a triaxial magnetometer 13 bit and a triaxial gyroscope 16 bit/axes with multiple sensitivity. This hardware is capable of acquiring and transmitting data to a computer through a Bluetooth connection and at the end of each analysis an automatic report containing the gait assessment results is ready to be analyzed.

SECONDARY OUTCOMES:
Posture | 10 minutes
  With this rating chart, postural changes that may occur in 13 different parts of the body are monitored and scored. The 13 body alignment segments include posterior views of the head, shoulders, spine, hip, feet, and arches, and lateral (left side) views of the neck, chest, shoulders, upper back, trunk, abdomen, and lower back. In this original version, each body segment was scored 5 (correct posture), 3 (slight deviation), or 1 (pronounced deviation). The total score obtained at the end of the test is maximum 65 and minimum 13
Pain Level | 1 minutes
  The Visual Analog Scale (VAS) pain score is a simple and effective method used to measure patients' pain levels. This method is typically represented by a line ranging from 0 to 10, where 0 indicates no pain and 10 indicates the most severe pain. Patients are asked to mark a point on the line that corresponds to their level of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Halil Ibrahim Bulguroglu, Study Director — Ankara Medipol University
Locations (1):
- Ankara Medipol University, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No